CLINICAL TRIAL: NCT07368504
Title: Development and Clinical Validation of an Artificial Intelligence-Based Interpretation System for Newborn Screening of Inherited Metabolic Disorders
Brief Title: AI for Newborn Metabolic Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, huzhenzhen, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2025-IRB-0550-P-01
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Inherited Metabolic Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI and Manual Interpretation of Newborn Screening Data (Other)
  Interventions: Diagnostic Test: Artificial intelligence-based interpretation system for newborn genetic metabolic disease screening

INTERVENTIONS:
Diagnostic Test: Artificial intelligence-based interpretation system for newborn genetic metabolic disease screening — This intervention is a deep learning-based software algorithm designed specifically for the interpretation of tandem mass spectrometry (MS/MS) data from routine newborn screening in Chinese neonates. It integrates clinical covariates-including gestational age, birth weight, and blood collection time-to perform multiple-of-the-median (MOM) normalization and simultaneously evaluates 42 inherited metabolic disorders. Unlike existing AI tools developed for older-generation screening panels (e.g., those covering only 29 analytes), this system is trained and validated on over 300,000 real-world Chinese newborn samples, making it the first AI diagnostic tool tailored to China's current expanded newborn screening program.

SUMMARY:
The goal of this clinical trial is to evaluate whether an artificial intelligence (AI)-based interpretation system can accurately diagnose inherited metabolic disorders in newborns undergoing routine screening. The main questions it aims to answer are:

What is the sensitivity and specificity of the AI system compared to standard manual interpretation? Does the AI system reduce variability in screening results? Researchers will compare the AI interpretation results with those from standard manual review by trained laboratory staff to assess diagnostic performance.

Participants will:

Have their routine newborn screening blood samples analyzed using both the AI system and standard manual interpretation Be followed according to national newborn screening guidelines if either method indicates a positive result

ELIGIBILITY:
Inclusion Criteria:

* Newborns who underwent routine newborn screening for inherited metabolic disorders at the Zhejiang Provincial Newborn Screening Center between May 2025 and December 2027
* Blood samples collected between 2 and 28 days of age
* Availability of complete newborn screening test data and essential clinical information

Exclusion Criteria:

* Missing, incomplete, or poor-quality screening data
* Duplicate samples from the same newborn

Ages: 2 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200000 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the AI interpretation system for detecting inherited metabolic disorders | Within 12 months after newborn screening
Specificity of the AI interpretation system for detecting inherited metabolic disorders | Within 12 months after newborn screening

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China